CLINICAL TRIAL: NCT05602766
Title: Ngenla® Subcutaneous Injection Special Investigation
Brief Title: Ngenla Subcutaneous Injection Special Investigation
Status: Active, not recruiting | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C0311011
Record Dates: First submitted 2022-10-27; First posted 2022-11-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-10

CONDITIONS: Growth Hormone Deficiency Without Epiphyseal Closure
Keywords: Growth hormone deficiency (GHD); Recombinant human growth hormone (hGH); once-weekly injection; Somatrogon
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — somatrogon

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- NGENLA (Somatrogon): Patients with GHD without epiphyseal closure who received NGENLA (Somatrogon)
  Interventions: Drug: NGENLA (Somatrogon)

INTERVENTIONS:
Drug: NGENLA (Somatrogon) — Dosage, Frequency: Refer to the latest package insert.

SUMMARY:
The purpose of this study is to learn about the long-term safety and effects of Ngenla. Ngenla is approved for treatment of GHD (Growth hormone deficiency) without epiphyseal closure under daily medical practice.

Registration criteria of this study are the patients who:

* Have GHD without epiphyseal closure and receiving Ngenla for the first time.
* Are boys less than 15 years or girls less than 13 years of age at the start of treatment with Ngenla.

All patients in this study will receive Ngenla according to the prescriptions. We will examine their experiences for a long time. This will help us to determine the safety and effects of Ngelna for long-term use.

Patients will be followed up from the date of first Ngenla treatment until November 30, 2027.

DETAILED DESCRIPTION:
This is a multi-center cohort study in patients with GHD without epiphyseal closure receiving NGENLA® Subcutaneous Injection. The investigators complete the case report form (CRF) based on the information extracted from the medical record created in daily medical practice.

ELIGIBILITY:
Patients who satisfy all of the registration criteria are subject to this study.

Registration criteria

1. Patients with GHD without epiphyseal closure who receive this drug for the first time after the date of contract for this study.
2. Boys who are less than 15 years and girls who are less than 13 years of chronological age at the start of treatment with this drug.

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients with GHD without epiphyseal closure who received NGENLA
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2023-02-06 (Actual); Primary Completion 2029-04-06 (Estimated); Study Completion 2029-04-06 (Estimated)

PRIMARY OUTCOMES:
The number of patients reporting Adverse Events (AEs) | up to 5 years
Incidence of Glucose metabolism disorders per exposure period | up to 5 years
Incidence of Neoplasm per exposure period | up to 5 years
Annual growth rate (cm/year) | up to 5 years
Growth rate standard deviation score (SDS) for chronological age | up to 5 years
Change in height SDS for chronological age and time-course of height SDS for chronological age | up to 5 years
Proportion of reported Adverse Events | up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C0311011